CLINICAL TRIAL: NCT00640692
Title: Kinase Genotyping of Gastrointestinal Stromal Tumors (GIST) From Patients Enrolled in the A6181112 Phase IIIb Trial at Participating U.S. and Ex-U.S. Medical Centers
Brief Title: Kinase Genotyping of Gastro Intestinal Stomach Tumors (GISTs) From Patients Enrolled in Pfizer A6181112 Phase IIIb Trial
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient enrollment
Sponsor: Oregon Health and Science University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Pfizer GIST Genotyping Study
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Gastrointestinal Neoplasm
Keywords: Gastrointestinal stromal tumor; GIST; Sunitinib; Imatinib
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genomic DNA from tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
The purpose of this study is to determine the genetic makeup of gastro intestinal stomach tumors (GISTs) from patients enrolled in the A6181112 phase IIIb trial. Tumor samples will be screened for mutations and this information will be used to determine whether the progression-free survival of patients being treated with the cancer medication sunitinib is related to the underlying genotype of their GIST.

DETAILED DESCRIPTION:
In this companion study, we will analyze the genomic DNA from the GIST tumor specimens of patients enrolled in the in the A6181112 phase IIIb trial at participating U.S. and ex-U.S. medical centers. Specifically, GIST samples will be screened for mutations in KIT gene exons 9, 11, 13 and 17, and PDGFRA gene exons 12, 14 and 18, to determine the primary kinase genotype. Subset analyses will be performed and compared with the overall PFS rates observed in patients with primary and secondary imatinib resistance. Based on data from a previous phase I/II trial, our hypothesis is that patients with either primary or secondary imatinib resistance having a KIT exon 9-mutant or WT GIST will have a longer PFS when treated with sunitinib than patients with exon 11-mutant GIST. We further hypothesize that this difference will be observed among patients treated with high-dose imatinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in Pfizer A6181112

Exclusion Criteria:

* Patients who do not consent for analysis of their tumor in this companion study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in Pfizer A6181112
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Estimated); Study Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Corless, MD, PhD, Principal Investigator — Oregon Health and Science University

REFERENCES:
- See also: Pfizer A6181112 phase IIIb trial — http://www.clinicaltrials.gov/ct2/show/NCT00372567?term=a6181112&rank=2